CLINICAL TRIAL: NCT02903901
Title: Melatonin for Prevention of Post- Operative Delirium Pilot Study Protocol
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator found that a new study drug that is FDA approved would be superior to melatonin
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Muralidhara Rao, Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 206981
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-09

CONDITIONS: Delirium
Keywords: Delirium
MeSH Terms: conditions — Delirium | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Individuals who are randomized to the control arm will receive liquid placebo sublingually 60-90 minutes prior to surgery.
  Interventions: Drug: Placebo
- Melatonin (Active Comparator): Individuals who are randomized to the treatment arm will receive 10 mg liquid IR-SL melatonin 60-90 minutes prior to surgery
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — 10 mg liquid Melatonin IR-SL at 7 pm for 1 week
  Arms: Melatonin
Drug: Placebo — 10 mg liquid placebo at 7 pm for 1 week
  Arms: Placebo

SUMMARY:
To test the efficacy of melatonin compared to placebo in preventing post-operative delirium and reduction in intensity or duration of delirium in individuals 65 years of age and older who undergo orthopedic surgery after low energy lower extremity fractures (LELEF).

Biomarkers may play important roles in the detection, prediction and management of delirium especially in frail elderly individuals. Predictive biomarkers may help characterize an individual's susceptibility to delirium and thereby help specialized treatment, care and management of such individuals during their hospitalization. They may also help predict treatment response to a specific modality and help in selection of such modality. Recent studies performed in the UK and published in 2011 have measured plasma cholinesterase activity and determined that these levels were lower in patients who developed delirium compared with remaining subjects. Other studies have indicated that CRP may also have a role in delirium prediction as they have found that CRP measured on admission to an ICU had predictable changes that occurred within 24 hours that in turn were predictors of delirium. One the aims of the study is to compare the predictive and treatment response values of groups of biomarkers that have been hypothesized to be of predictive value.

DETAILED DESCRIPTION:
Surgery causes oxidative stress on the brain9 leading to inflammation. Post-operative delirium has been linked with inflammation in the brain. Delirium has been hypothesized to be a central nervous system response to systemic inflammation during a state of blood-brain barrier (BBB) compromise.

Studies have shown a rise of inflammatory cytokines and fall of anti-inflammatory cytokines. Vice-versa, external cytokine administration has been shown to lead to delirium. Melatonin is known for its strong anti-oxidant and anti-inflammatory properties, this should account for its preventive properties in post-operative delirium. It has also been hypothesized that post-operative delirium in elderly is caused by circadian rhythm disturbances secondary to a relative lack of melatonin.

Keeping in mind the above two possible pathophysiology for delirium, investigators are expecting melatonin supplementation should be able to reduce the incidence of post-operative delirium particularly in elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65 years of age and older undergoing Low Energy Lower Extremity Fractures (LELEF) surgery
* Presence of an LELEF fracture
* Low Energy (e.g., falls from standing height, falls from sitting, etc.).
* Operative Fractures:

  * Pathologic femur and tibia fractures
  * Femoral neck fractures
  * Pertroch: including intertroch, subtroch fractures
  * Femoral shaft
  * Supracondylar femur fractures
  * Periprosthetic fractures around total hip and total knee arthroplasties
  * Tibial plateau fractures
  * Proximal Tibia Fractures
  * Tibial Shaft Fractures
  * Distal 1/3 tibia fractures
  * Ankle Fractures that are admitted

Exclusion Criteria:

* Patients with previous adverse reaction or side-effects to melatonin
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.
* Inability to communicate in English
* Patients with a Montreal Cognitive Assessment (MoCA) score of below 7 will not be included in the study because of their inability to give informed consent at that stage. This score is approximately 2 standard deviation below average score for Alzheimer's Dementia.
* Participants who are unable to give consent or communicate well in English will not be enrolled

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Delirium assessment | 1 Week
  The Delirium Rating Scale Revised (DRS-R98) will be given to all patients every day for seven days. Investigators will compare the scores recorded on day 7 between those receiving melatonin versus those receiving placebo controlling for their baseline performance.

SECONDARY OUTCOMES:
Hospital stay | 1 Week
  Length of hospital stay will be recorded for all patients and compared between the two treatment groups (i.e., those receiving melatonin and those receiving placebo).

CONTACTS AND LOCATIONS:
Overall Officials: Muralidhara S Rao, MD, Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

REFERENCES:
- [Background] Deiner S, Silverstein JH. Postoperative delirium and cognitive dysfunction. Br J Anaesth. 2009 Dec;103 Suppl 1(Suppl 1):i41-46. doi: 10.1093/bja/aep291. PMID 20007989
- [Background] Bekker AY, Weeks EJ. Cognitive function after anaesthesia in the elderly. Best Pract Res Clin Anaesthesiol. 2003 Jun;17(2):259-72. doi: 10.1016/s1521-6896(03)00005-3. PMID 12817919